CLINICAL TRIAL: NCT02925780
Title: In Vivo Action of Infiltrating Resin Icon® on Fluorosis - a 12 Month Follow up Trial
Brief Title: 12 Month Follow up in Vivo Icon Study on Fluorotic Teeth
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Organisational and regulatory challenges.
Sponsor: DMG Dental Material Gesellschaft mbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIAFLUOR
Record Dates: First submitted 2016-09-28; First posted 2016-10-06 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Fluorosis; Oral Deseases
Keywords: Enamel defects; Fluorosis; Icon; Resin infiltration
MeSH Terms: conditions — Fluoride Poisoning | interventions — Enamel Microabrasion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resin infiltration (Experimental): The labial surface of fluorosed teeth (upper front teeth) that are selected for this group will be treated using the resin infiltrant "Icon" (DMG, Germany). This is a minimally invasive treatment to improve the aesthetics by masking the white spots.
  Interventions: Device: Resin infiltration
- Microabrasion (Active Comparator): The labial surface of fluorosed teeth (upper front teeth) that are selected for this group will be treated by microabrasion using the microabrasive material "Opalustre" (Ultradent, USA). This is a minimally invasive treatment to improve the aesthetics by masking the white spots.
  Interventions: Device: Microabrasion

INTERVENTIONS:
Device: Resin infiltration — Teeth selected for this group will be treated with the resin infiltrant Icon according to the manufacturer's instructions. In short, teeth will be isolated with a rubber dam and the labial tooth surface cleaned with non-fluoride prophylactic paste and pumice. After an etching and drying step (to open the lesion surface), Icon will be applied following the manufacturer's instructions and subsequently light cured, followed by polishing.
  Digital images are taken before and after the treatment as well as at the follow-up visits (3, 6, 9 and 12 months).
  Other Names: Icon (DMG, Germany), Approximal resin infiltration kit
  Arms: Resin infiltration
Device: Microabrasion — The labial surfaces of teeth selected for this group will be isolated and precleaned. Subsequently, the microabrasive material, Opalustre, will be applied according to the manufacturer's instructions, using a rubber cup at low speed (5 times each for 5 seconds). Between each of the applications the surface is washed by flushing water using a syringe.
  Digital images are taken before and after the treatment as well as at the follow-up visits (3, 6, 9 and 12 months).
  Other Names: Opalustre (Ultradent, USA)
  Arms: Microabrasion

SUMMARY:
Clinical trial to investigate the clinical efficiency of resin infiltration compared to microabrasion in the improvement of dental fluorosis.

DETAILED DESCRIPTION:
Dental fluorosis is an endemic public health concern that develops if infants are subjected to excessive amounts of fluoride during enamel formation. Anatomopathologically, dental fluorosis presents itself as a hypermineralized surface layer and subsurface hypomineralization involving the external third of the thickness of the enamel, which is equivalent to early carious lesions. In addition, fluorosis features a number of clinical changes in the enamel surface, ranging from the appearance of thin white lines up to severe structural defects, thereby compromising overall esthetics, which sometimes leads to children dropping out of school due to its psychological impact.

The aim of this controlled clinical trial is to evaluate the efficacy of enamel microabrasion and resin infiltration in improving the dental esthetic of patients with fluorosis. Resin infiltration is a microinvasive technique that can improve the esthetics by infiltrating a low-viscosity resin (that has a similar refractive index to enamel) into the porose hypomineralized enamel of fluorosed white spots. This approach thus largely preserves the enamel compared to more invasive techniques such as microabrasion and has been shown to be efficient in previous studies.

This study will be conducted in the provinces of Pichincha and Cotopaxi, Ecuador and patients between 10 to 12 years of age with stage 1, 2, and 3 fluorosis according to the Thylstrup and Fejerskov (TF) scale or questionable, very mild, and mild fluorosis according to Dean's Index will be recruited. In addition to the immediate esthetic improvement, long term stability of the outcome will be assessed at 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Questionable, Very mild, and Mild (Dean's Index) dental fluorosis as well as TF scale grades 1, 2, and 3 of the upper anterior teeth.
* Parents of children who accept and commit to the informed consent letter collaborate with the study taking their children to each of the scheduled follow ups.

Exclusion Criteria:

* Teeth without fluorosis.
* Teeth with hypoplasia.
* Teeth with incipient caries lesions observed at gingival level and differentiated by the Presence of plaque.
* Teeth previously restored or with aesthetic corrective treatments
* Teeth with endodontic treatment.
* Patients with low or questionable hygiene.
* Malnourished patients or that have some underlying disease.
* Teeth with less than two thirds of its visible crown.
* Children that have less than six teeth in their oral cavity.
* Allergic reaction to methylmethacrylate.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
action of DMG Icon-infiltrative ® resin and micro abrasion to mask fluorotic enamel | immediate after treatment
  Evaluate the action of DMG Icon-infiltrative resin and micro abrasion immediately after application to mask fluorotic teeth by comparison of pre- vs. post-treatment photographs

SECONDARY OUTCOMES:
Surface changes | 12 month
  changes that occur on the surface of the teeth with fluorosis, which have been treated with DMG Icon ® and micro-abrasion assessed via photographs
Clinical characteristics Icon | 3, 6, 9, 12 month
  clinical characteristics of the tooth surfaces that have been treated with DMG Icon ® and micro-abrasion and its relationship to the degree of fluorosis
Efficacy of infiltration to mask fluorotic teeth long-time | 12 month
  Compare the benefit of the infiltrative resin DMG Icon related to micro abrasion Opalustre ULTRADENT as control procedure, focus: stabilisation of masking quantified by photographs

CONTACTS AND LOCATIONS:
Overall Officials: Ana Armas Vega, Principal Investigator — Universidad Internacional del Ecuador

IPD SHARING:
Plan to Share IPD: No